CLINICAL TRIAL: NCT03826537
Title: An Open-label, Non-randomised Study to Investigate the Pharmacokinetics of Tutin and Hyenanchin, Following Single Dose Administration of Honey Containing Tutin and Hyenanchin to Healthy Male Subjects
Brief Title: A Study of How Tutin and Hyenanchin, Two Toxins Found in Honey, Are Absorbed and Processed by the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christchurch Clinical Studies Trust Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CH-1101; NCT01531556 (obsolete NCT alias)
Record Dates: First submitted 2012-08-05; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Tutin Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Honey substance (Other): Honey substance containing 5.1 mg/kg tutin and 23 mg/kg hyenanchin. Subjects to receive single dose of test material such that each subject receives 1.8 mcg/kg body weight of tutin.
  Interventions: Other: Honey substance

INTERVENTIONS:
Other: Honey substance — Honey substance containing 5.1 mg/kg tutin and 23 mg/kg hyenanchin

SUMMARY:
Honey available in New Zeland can contain the toxins tutin and hyenanchin. Tutin is produced by several plants native to New Zealand. Bees collect honeydew contaminated with tutin and hyenanchin for honey production.

Honey contaminated with high levels of tutin has caused cases of poisoning in New Zealand since the 1800s, with the most recent outbreak in 2008.

The study aims to find out how tutin and hyenanchin are absorbed and processed by the body. This information will help the FSANZ give guidance on acceptable levels of tutin and hyenanchin in honey.

About 6 healthy men will each take a single dose of honey containing known concentrations of tutin and hyenanchin.

This dose level is similar to what someone who eats a lot of honey would have, if the honey contained the maximum level of tutin allowed under the Food Standards Code.

Blood tests to measure tutin and hyenanchin levels will be taken at certain times after dosing, and any side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, aged between 18 and 55 years, inclusive.
2. Healthy on the basis of medical history and screening assessments.
3. Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive.
4. Agree to abstain from alcohol consumption from 48 hours before dosing through to the completion of pharmacokinetic samples.
5. Able to participate, and willing to give written informed consent and to comply with the study protocol requirements.

Exclusion Criteria:

1. A history of clinically relevant cardiovascular, gastrointestinal, hepatic, renal,endocrine, pulmonary, neurological, psychiatric, allergic or skin disorders.
2. Any gastrointestinal condition, disorder or previous surgery that, in the opinion of the investigator, may interfere with absorption of study product.
3. History of or symptoms suggestive of significant gastro-esophageal reflux disease or peptic ulcer disease.
4. Significant neurological history, including relevant history of seizure disorders, major head trauma or cerebrovascular disease.
5. Known allergy or hypersensitivity to honey.
6. Sustained blood pressure levels at screening of < 90 mmHg or > 150 mmHg for SBP or < 50 mmHg or >90 mmHg for DBP.
7. Sustained resting heart rate (HR) > 100 or < 40 beats per minute (bpm) at screening.
8. Clinically significant abnormalities in laboratory test results at screening or baseline.
9. Positive serology screen for HIV, or Hepatitis B or C at screening.
10. Positive results on urine drug / alcohol test at screening or Day 1 (if performed).
11. Smokers of >10 cigarettes/day within 3 months prior to admission and unable to stop smoking during the study.
12. Participation in an investigational drug study within 1 month prior to dosing.
13. Blood or plasma donation of > 500 mL within the 3 months prior to dosing.
14. Prescription or herbal remedies taken within 7 days or 5 half-lives (whichever is longer) prior to dosing. Over-the-counter medications and vitamins are not permitted within 72 hours prior to dosing. Paracetamol is permitted as required throughout the study, to a maximum of 4 grams per day.
15. Consumption of food or beverages containing honey within 72 hours prior to dosing.
16. Known or suspected previous tutin poisoning.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of tutin and hyenanchin (Tmax) | Pre-dose through to 24 hours post dose. May be modified according to sentinal PK results.
  Time to maximum plasma concentration (Tmax)
Pharmacokinetics of tutin and hyenanchin (AUC) | Pre-dose through to 24 hours post dose
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics of tutin and hyenanchin (Cmax) | Pre-dose through to 24 hours post dose
  Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wynne, MBChB, Principal Investigator — Christchurch Clinical Studies Trust
Locations (1):
- Christchurch Clinical Studies Trust, Christchurch, Canterbury, New Zealand